CLINICAL TRIAL: NCT03649295
Title: Randomized Study of the Influence of Functional Electrical Stimulation in Patients With Dysphagia After Stroke
Brief Title: Combined Conventional Speech Therapy and Functional Electrical Stimulation in Dysphagia Following Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Geral de Fortaleza (Other Government)
Responsible Party: Principal Investigator, Klayne Cunha Matos, Principal Investigator, Hospital Geral de Fortaleza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2388931
Record Dates: First submitted 2018-08-21; First posted 2018-08-28 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Dysphagia, Oropharyngeal; Stroke, Ischemic
MeSH Terms: conditions — Deglutition Disorders; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Electrical Stimulation (Experimental): - Functional electrical stimulation device obeying the following steps: Muscle heating - 2 min, 10 Hz, 250 μm; Potentiation of muscle fibers type I - 8 min, 30 Hz, 250 μm; Potentiation of muscle fibers type II - 8 min, 80 Hz, 300 μm; Toning - 8 min, 30 Hz, 300 μm; Muscle Relaxation - 4 min, 5 Hz, 200 μm One channel of electrodes will be placed in the submental region and the other in the thyroid. Treatment should be started at minimum levels of intensity, increasing carefully until appropriate effects are achieved in the procedure. Conventional therapy should be performed in conjunction with functional electrostimulation
  -Conventional speech therapy with laryngeal elevation exercises, stimulation of oral reflexes, tongue movements, lips and cheeks, gustatory therapy
  Interventions: Other: Functional Electrical Stimulation; Other: Conventional Speech Therapy
- Placebo (Placebo Comparator): Sham.The electrodes are placed at 0 Hz
  -Conventional speech therapy with laryngeal elevation exercises, stimulation of oral reflexes, tongue movements, lips and cheeks, gustatory therapy
  Interventions: Other: Conventional Speech Therapy

INTERVENTIONS:
Other: Functional Electrical Stimulation — Functional electrical stimulation device obeying the following steps:
  Muscle heating - 2 min, 10 Hz, 250 μm; Potentiation of muscle fibers type I - 8 min, 30 Hz, 250 μm; Potentiation of muscle fibers type II - 8 min, 80 Hz, 300 μm; Toning - 8 min, 30 Hz, 300 μm; Muscle Relaxation - 4 min, 5 Hz, 200 μm One channel of electrodes will be placed in the submental region and the other in the thyroid. Treatment should be started at minimum levels of intensity, increasing carefully until appropriate effects are achieved in the procedure
  Arms: Functional Electrical Stimulation
Other: Conventional Speech Therapy — Conventional speech therapy with laryngeal elevation exercises, stimulation of oral reflexes such as swallowing reflex, tongue movements, lips and cheeks, gustatory therapy

SUMMARY:
This study will evaluate the effectiveness of conventional speech therapy associated with functional electrical stimulation in patients with dysphagia after ischemic stroke. Included patients will be divided into two groups, where in the intervention group the speech therapy is associated to functional electrical stimulation, and in the control group, the patients will receive the conventional speech therapy with electrical stimulation Placebo with intensity 0hz.

DETAILED DESCRIPTION:
Since the 1980's, electrical stimulation has been used for therapeutic purposes in Brazil, and, since 1990's, it has been used as a relevant therapeutic tool in the cases of oropharyngeal dysphagia in addition to speech therapy. Positive results have been observed in the treatment of swallowing disorders, including in patients that carry neurological diseases. However, there is no substantial evidences for this interventions.

In this study, the electrotherapy will be used as a complement to conventional speech therapy and performed the application of electrical stimulation protocol in dysphagia, through the apparatus Neurodyn Portable TENS/FES (transcutaneous electrical neurostimulation/ functional electrical stimulation), which is a transcutaneous neuromuscular stimulator flow TENS/FES from two channels with independent intensity adjustment. It is about a non-invasive technique with no systemic effect, causing no dependence or undesirable side effects, and consists by gentle application in electrical stimulation, through electrodes placed in body areas affected by pain or to activate skeletal muscles and produce movements. A channel of electrodes will be placed in the submental region and the other channel on the thyroid cartilage., in formation of a T. The explication of the procedure in the patient treatment, is describing the sensations that he should expect that happened during the stimulation. The intensity of necessary flow to apply in the treatment, will depend in the sensation of the patient, therefore, it is applicable until the tolerance level or desirable muscular contraction. Thus, the treatment should be initiated with minimal levels of intensity, by being carefully raised if appropriate effects are achieved on the procedure and according to the patient report.

ELIGIBILITY:
Inclusion Criteria:

* Stroke - ischemic type;
* Dysphagia following stroke;
* 40 to 70 years old;
* Exclusive enteral Feeding;
* Glasgow > 11.

Exclusion Criteria:

* Pregnants;
* Febrile Condition;
* Neoplasia;
* Pacemaker;
* Cochlear Implant;
* Anxious Patient;
* Degenerative Neurological Diseases.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-07-26 (Actual); Study Completion 2020-07-26 (Actual)

PRIMARY OUTCOMES:
Level of dysphagia assessed by videoendoscopy of swallowing | 5 days ( before and immediately after intervention)
  Anatomical Evaluation:Tongue, palate, pharynx, larynx - normal or specify changes
  Functional Evaluation:
  * Mobility (lips/tongue), tongue's sensitivity, palatine veil's closure - adequate or inadequate
  * Pharynx - salivary/alimentary stasis
  * Larynx - normal, decreased mobility, unilateral or bilateral immobility
  Deglutition assessment (liquid, thick, pasty and solid foods):
  -Delay of swallowing, anterior/posterior escape, stasis in vallecula/pyriform sinuses, laryngeal penetration, laryngotracheal aspiration - present or absent
  Functional swallowing: alteration in anatomical or functional evaluation with absence of salivary/alimentary stasis Mild dysphagia: there is also salivary or food stasis in only one consistency with efficient maneuvers such as lowered head, Masako or effortless swallowing Moderate dysphagia: there is also laryngeal penetration to one or more consistencies Severe dysphagia: there is also laryngotracheal aspiration or absence of swallowing reflex
Safe food Intake assessed by Functional Scale Oral Ingestion - FOIS | 5 days (before and immediately after intervention)
  Measured by the Functional Oral Ingestion Scale (FOIS). FOIS results are rated on a scale of 1 to 7 levels. The levels will increase according to the safe amount of oral diet ingested by the patient safely.
  Level1 - nothing by mouth; Level 2 - tube dependent with minimal attempts of Food or liquid; Level 3 - tube dependent with consistence oral Intake of Food or liquid; Level 4 - total oral diet of a single consistency; Level 5 - total oral diet with multiple consistencies but requiring special preparation or compensations; Level 6 - total oral diet with multiplex consistencies without special preparation, but with specific Food limitations; Level 7 - total oral diet with no restrictions.

SECONDARY OUTCOMES:
Clinical evaluation of swallowing through the risk assessment protocol for dysphagia - PARD | 5 days (before and immediately after intervention)
  Before feeding:
  * Comprehensive language, oral reflexes(vomiting, trismus, deglutition) and sialorrhea- present or absent
  * Inside oral and facial sensitivity- present or reduced
  During feeding (liquid, thick and pasty):
  * Captation, anterior and posterior escape, cough reflex and gagging- present or absent
  * Oral transit time, number of swallowing, laryngeal elevation- adequate or inadequate
  * Voice normal or "wet"
  Functional swallowing- there are changes that do not compromise safe feeding as reduced sensitivity (intra-oral or facial), anterior escape due to small anatomical or functional changes Mild dysphagia- multiple swallowing, inadequate laryngeal elevation, "wet" voice but cough reflex efficient Moderate dysphagia- multiple swallowing, inadequate laryngeal elevation, "wet" voice, weak cough reflex and gagging one or more consistencies Severe dysphagia- when there is no evidence of coughing, swallowing reflexes or gagging difficult to recover

CONTACTS AND LOCATIONS:
Overall Officials: Klayne C Matos, MD, Principal Investigator — Hospital Geral de Fortaleza
Locations (1):
- Ubiversidade Federal do Ceará, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Turn the study public to contribute to the science around the world, by publishing results and share knowledge to future researchers.

REFERENCES:
- [Derived] Matos KC, de Oliveira VF, de Oliveira PLC, Carvalho FA, de Mesquita MRM, da Silva Queiroz CG, Marques LM, Lima DLN, Carvalho FMM, Braga-Neto P. Combined conventional speech therapy and functional electrical stimulation in acute stroke patients with dyphagia: a randomized controlled trial. BMC Neurol. 2022 Jun 22;22(1):231. doi: 10.1186/s12883-022-02753-8. PMID 35733098